CLINICAL TRIAL: NCT06479291
Title: The Efficacy and Safety of Hydroxychloroquine Plus TPO-RA in Antinuclear Antibody-positive Patients With Primary Immune Thrombocytopenia-- The Multicenter, Randomized, Open-labled Clinical Trial
Brief Title: The Efficacy and Safety of HCQ Plus TPO-RA in ANA Positive ITP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunfeng Cheng (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai Jinshan Hospital (Other); Zhongshan Qingpu Hospital, Fudan University (Unknown); Zhongshan Wusong Hospital, Fudan University (Unknown); Macau University of Science and Technology Hospital (Other); Health and Humanity Research Centre, Hongkong (Unknown); Dr. Stanley Ho Medical Foundation, Macau (Unknown)
Responsible Party: Sponsor-Investigator, Yunfeng Cheng, Professor of Institute of Clinical Science, Zhongshan Hospital, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2024-027R2
Record Dates: First submitted 2024-06-22; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Immune Thrombocytopenia With Positive ANA Antibodies
MeSH Terms: interventions — Hydroxychloroquine; eltrombopag

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCQ plus TPO-RA group (Experimental): This group is experiment group. Participants will take eltrombopag for at least 24 weeks, the dose of eltrombopag is adjusted according to participants' platelet count, with HCQ twice a day for 1 year
  Interventions: Drug: Hydroxychloroquine Oral Tablet; Drug: Eltrombopag
- TPO-RA group (Placebo Comparator): This group is control group. Participants will take eltrombopag for at least 24 weeks, the dose of eltrombopag is adjusted according to participants' platelet count.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Hydroxychloroquine Oral Tablet — Hydroxychloroquine is taken at the dose of 0.1g / dose, twice a day for 1 year, regardless of food intake.
  Other Names: Hydroxychloroquine
  Arms: HCQ plus TPO-RA group
Drug: Eltrombopag — Participants will take eltrombopag for at least 24 weeks, the dose of eltrombopag is adjusted according to participants' platelet count.
  Other Names: Eltrombopag pill

SUMMARY:
The goal of this clinical trial is to learn if hydroxychloroquine (HCQ) plus thrombopoietin receptor agonists (TPO-RA) works to treat primary immune thrombocytopenia with positive anti-nuclear antibodies in adults. It will also learn about the safety of HCQ plus TPO-RA. The main questions it aims to answer are:

Does HCQ plus TPO-RA raise the response rate in participants, compared to TPO-RA alone? Does HCQ plus TPO-RA prolong the response duration in participants, compared to Pred alone? Does HCQ plus TPO-RA decrease the dose of TPO-RA to maintain response in participants, compared to TPO-RA alone? What medical problems do participants have when taking HCQ plus TPO-RA? Researchers will compare HCQ plus TPO-RA with TPO-RA alone to see if HCQ plus TPO-RA works better to treat primary immune thrombocytopenia with positive anti-nuclear antibodies.

Participants will:

Take TPO-RA every day for no more than 24 weeks, adjust the dose of TPO-RA according to the platelet level, with or without HCQ twice a day for 1 year; Visit the clinic once every 1 weeks for the first 8 weeks, and once every 2-4 weeks in the following 10 months for checkups and tests; Keep a diary of their symptoms

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (Primary immune thrombocytopenia, ITP) is an acquired autoimmune hemorrhagic disease characterized by a decreased peripheral platelet count and an increased risk of bleeding. It has been reported that 33.3% -39.2% of ITP patients have positive antinuclear antibodies (ANA) in the course of the disease.In the meantime, they do not meet the diagnostic criteria for rheumatic diseases such as lupus erythematosus(SLE). ITP patients with positive ANA are prone to relapse and chronicity. Therefore, it is necessary to explore new clinical treatments to attain long-term remission in these patients.

Hydroxychloroquine (HCQ) has immune modulating role on a variety of immune cells.A clinical trial enrolled immune thrombocytopenia secondary to SLE, and ITP with positive anti-nuclear antibodiy (ANA) were treated with HCQ combined with glucocorticoids. The results showed an overall response rate of 60% (24 / 40), including 18 continuous complete response (CR) and 6 continuous response (R), and some patients had continued elevated platelet counts 3 months after treatment initiation. The above studies illustrate that HCQ contributes to the treatment of chronic ITP, especially as a long-term therapeutic agent with low economic burden and good tolerance. In patients who do not response to HCQ plus corticosteroids, TPO-RA, a second line treatment, will be recommended. By now, no study has assess the efficacy and safety of HCQ plus TPO-RA in these patients. In the current study, the question will be answered.

ELIGIBILITY:
Inclusion Criteria:

1. Age is above 15 years old.
2. Before randomization, the clinical diagnosis is primary immune thrombocytopenia. The platelet count is less than 30×10^9 / L within 1 week before enrollment, or platelet count is less than 50×10^9 / L with bleeding symptoms within 1 week before enrollment.
3. The antinuclear antibody is positive.
4. Other autoantibodies (mainly including dsDNA antibodies, SSA, SSB, RNP, β 2-GP, ACA, ANCA) are negative.
5. Participants who had received at least two HD-DXM 40 mg/d ×4 d, failed or relapsed, or received standard dose prednisone (1-2 mg/kg/d) for 4 weeks, the platelet count remained <30×10 9 / L, or the platelet count normalized but decreased with prednisone tappering off, or prednisone 30mg to maintain the platelet number.
6. Prothrombin time does not exceed ± 3s of the normal value ranget, activated partial thrombin time is not outside normal range ± 10s; no history of coagulopathy except ITP.

(6)Understand the study procedures and sign the written informed consent form.

Exclusion Criteria:

1. Secondary thrombocytopenia caused by myelodysplastic syndrome, immune diseases such as systemic lupus erythematosus, early aplastic anemia, atypical reanemia, antiphospholipid syndrome, thrombotic thrombocytopenic purpura and various other causes.
2. The participant has experienced any arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), or clinical symptoms and medical history indicate thrombophilia.
3. Congestive heart disease, including New York Heart Association (NHYA) Grade III / IV, occurred within 3 months prior to screening, arrhythmia requiring medication or myocardial infarction, or arrhythmia known to increase the risk of thrombotic events (such as atrial fibrillation), or corrected QT interval (QTc) is longer than 450 ms, or QTc> 480 ms in paricipants with bundle branch block.
4. A medical history of parenchymal organ transplantation or allogeneic bone marrow transplantation.
5. Having received any medication affecting platelet function ( Including but not limited to aspirin, aspirin-containing complexes, clopidogrel, salicylates, and / or non-steroidal anti-inflammatory drugs NSAIDs ) or anticoagulant therapy for over consecutive 3 days within 2 weeks before screening.
6. With Glucose-6-phosphate dehydrogenase deficiency.
7. With retinal or visual field changes caused by 4-aminoquinoline compounds.
8. Being allergic to 4-aminoquinoline compounds.
9. Having evidence of Human Immunodeficiency Virus (HIV)/ hepatitis C virus(HCV)/ hepatitis B virus(HBV) infection (HIV antibody or HCV antibody is positive, HBV surface antigen is positive, or HBV surface antigen is negative but HBV-DNA indicating viral replication.
10. Glutamate transaminotransferase (ALT) or glutamate transaminase (AST) is higher than 1.5 times the upper limit of normal value (ULN), or total bilirubin or blood creatinine is higher than 1.2 times the ULN.
11. With liver cirrhosis or portal hypertension.
12. With evidence of malignant tumor activity, or receiving anti-tumor treatment within 5 years prior to the screening.
13. Participants being pregnant or lactating, or with potential fertility, reluctance to use effective contraception within the entire trial cycle and within 28 days after the end of the trial (or within 28 days after premature withdraw).

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 4 weeks
  The percentage of participants with platelet counts higher than 30×10^9/L and at least twice the baseline platelet count , for at least two consecutive tests (7 days apart).

SECONDARY OUTCOMES:
Complete response rate | 1 year
  The percentage of participants with platelet counts higher than 100×10^9/L , for at least two consecutive tests (7 days apart).
Duration of response | 1 year
  Time from response to disease relapse (platelet count ≤ 30×10^9/L on any test or occurance of bleeding symptoms )
Durable response rate | 1 year
  Percentage of patients with complete remission lasting at least 6 months without any additional ITP-specific therapy
Platelet count at each visit | 1 year
  Average platelet count at each visit
Time to response | 4 weeks
  Time from starting treatment to response
Time to TPO-RA withdrawal | 24 weeks
  Time from starting treatment to TPO-RA withdrawal
Rate of TPO-RA withdrawal | 24 weeks
  Rate of participants who withdraw TPO-RA with platelet count over 30×10^9/L
The maximum dose of TPO-RA to attain response | 8 weeks
  The maximum dose of TPO-RA to attain response (platelet count over 30×10^9/L)
Response rate throughout the trial | 1 year
  The percentage of response participants (platelet counts higher than 30×10^9/L and at least twice the baseline platelet count ) at each visit
Once response rate throughout the trial | 1 year
  The percentage of once response participants (platelet counts higher than 30×10^9/L and over twice the baseline platelet count for at least one visit) throughout 1 year
WHO bleeding score | 1 year
  WHO bleeding score at each visit
Adverse reaction | 1 year
  Adverse reaction at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Yunfeng Cheng, Principal Investigator — Shanghai Zhongshan Hospital
Locations (7):
- China (4):
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Wusong Hospital, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Jinshan Hospital, Shanghai, Shanghai Municipality
  - Qingpu Branch of Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
- Health and Humanity Research Centre, Hongkong, China., Hong Kong, Hong Kong
- Macau (2):
  - Dr. Stanley Ho Medical Foundation, Macao
  - University Hospital, Macau University of Science and Technology., Macao

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD information will become available starting 6 months after publication, for 1 year.

REFERENCES:
- [Background] Neunert C, Terrell DR, Arnold DM, Buchanan G, Cines DB, Cooper N, Cuker A, Despotovic JM, George JN, Grace RF, Kuhne T, Kuter DJ, Lim W, McCrae KR, Pruitt B, Shimanek H, Vesely SK. American Society of Hematology 2019 guidelines for immune thrombocytopenia. Blood Adv. 2019 Dec 10;3(23):3829-3866. doi: 10.1182/bloodadvances.2019000966. PMID 31794604
- [Result] Khellaf M, Chabrol A, Mahevas M, Roudot-Thoraval F, Limal N, Languille L, Bierling P, Michel M, Godeau B. Hydroxychloroquine is a good second-line treatment for adults with immune thrombocytopenia and positive antinuclear antibodies. Am J Hematol. 2014 Feb;89(2):194-8. doi: 10.1002/ajh.23609. Epub 2013 Nov 20. PMID 24254965
- [Result] Mejdoub S, Hachicha H, Gargouri L, Feki S, Mahfoudh A, Masmoudi H. Antinuclear antibodies in children: clinical signification and diagnosis utility. Tunis Med. 2021 Octobre;99(10):980-984. PMID 35288899
- [Result] Lambert MP, Gernsheimer TB. Clinical updates in adult immune thrombocytopenia. Blood. 2017 May 25;129(21):2829-2835. doi: 10.1182/blood-2017-03-754119. Epub 2017 Apr 17. PMID 28416506